CLINICAL TRIAL: NCT04624061
Title: Leveraging the HIV Platform for Hypertension Control in Uganda
Brief Title: Leveraging the HIV Platform for Hypertension Control in Uganda (INTEGRATED HIV/HTN) STUDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Infectious Diseases Research Collaboration, Uganda (Other)
Collaborators: Makerere University (Other); Uganda Heart Institute (Other); Ministry of Health, Uganda (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-156; 22196 (Other: London School of Hygiene and Tropical Medicine)
Record Dates: First submitted 2020-10-27; First posted 2020-11-10 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-07

CONDITIONS: HIV; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The integrated HIV/HTN care model with the following components;
  1. Training and capacity building on the INTEGRATED HIV/HTN model and NCD care
  2. Integrated HIV/HTN care delivery model by promoting HTN screening and care in HIV clinics.
  3. HMIS enhancements through mentorship and coaching on the use of NCD registers and NCD patient cards and HTN data capture in the (Electronic Medical Record) EMR system.
  4. SMS and/or WhatsApp for data coordination and communication among providers, District Health officers (DHOs) and study team (Mentors) to strengthen feedback.
  Interventions: Behavioral: Integrated HIV/HTN care model
- Control (No Intervention): Standard of care maintained. These are procedures conducted during the routine HIV and Hypertension care visits at the health facilities include;a) Provision of BP machines b)Provision of NCD register and NCD patient card and ; c) Following MOH treatment guidelines

INTERVENTIONS:
Behavioral: Integrated HIV/HTN care model — The intervention is a multi-component intervention of combined HIV and HTN care, based on the PRECEDE framework, to continuously identify barriers and facilitators leads to better health outcomes including dual control of HIV/HTN among adults in HIV care in the intervention compared to control facilities
  Arms: Intervention

SUMMARY:
The INTEGRATED HIV/HTN is a hybrid type-1 effectiveness/implementation cluster randomised trial evaluating the introduction of a multi-component integrated HIV/HTN care model intervention, randomised to 13 districts in the intervention arm compared to 13 districts in the control. Selected health facilities within the 13 intervention districts will receive the intervention while those in the 13 control districts will continue implementing the standard of care as per the Ministry of Health (MoH) guidelines. All the participating facilities will receive blood pressure (BP) machines, and Non- communicable diseases (NCDs) registers as a standard of care.

DETAILED DESCRIPTION:
The investigators propose to evaluate a multi-component integrated HIV/HTN care intervention through a cluster randomised controlled trial. A cluster has been defined at the level of the district which is the randomisation unit. A total of 26 districts will be randomised. Selected health facilities within the 13 intervention districts will receive the multi-component intervention of combined HIV and (hypertension) HTN care which includes; 1) Training and capacity building on the INTEGRATED HIV/HTN model and NCD care; 2) the Integrated HIV/HTN care delivery model by promoting HTN screening and care in HIV clinics; 3) Health management information system (HMIS) enhancements through mentorship and coaching on the use of NCD registers and NCD patient cards and HTN data capture in the EMR system; and 4) Short messaging system (SMS) and/or WhatsApp for data coordination and communication among providers, DHOs and the study team (who acts as mentors). The 13 control districts will continue implementing the current standard of care as per MoH guidelines.

The investigators will test the hypothesis that a multi-component intervention of combined HIV and HTN care, based on the PRECEDE framework, to continuously identify barriers and facilitators leads to better health outcomes including dual control of HIV/HTN among adults in HIV care in the intervention compared to control facilities.

Specific Objectives are as follows;

1. To determine the effectiveness of an integrated HIV/HTN care model on HTN and dual HIV/HTN control among adult patients in HIV clinics.
2. To assess the barriers and facilitators of the integrated HIV/HTN care model for HIV patients at different levels.
3. To determine the cost, cost-effectiveness and incremental gain costs of the integrated HIV/Hypertension care model approach.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and above with HIV for one category
* Adults 18 years and above with HIV and hypertension for the second category
* Willing to consent

Exclusion Criteria:

* Patients who are very sick
* Patients not willing to continue seeking care from the study health facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV patients screened for Hypertension(HTN) at Month 24 | Month 24
  Proportion of HIV patients Screened for HTN at 24 months months of follow up
Proportion of HTN patients diagnosed and started on treatment | Month 24
  Proportion of HTN patients diagnosed and started on treatment
Proportion of HIV/HTN patients with HTN Control (systolic blood pressure below 140 mm Hg and diastolic blood pressure below 90 mm Hg) at 12 months and 24 months. | 24 months
  Proportion of HIV infected patients with with documented history of elevated blood pressure or prior HTN diagnosis on medication who are controlled (systolic blood pressure below 140 mm Hg and diastolic blood pressure below 90 mm Hg) at 12 months and 24 months.
Proportion of HIV/HTN patients with HIV/HTN Dual Control: (who are both "HTN controlled" and have undetectable HIV viral load (at 12 months and 24 months). | 24 months
  Proportion of HIV/HTN patients with HIV/HTN Dual Control: (who are both "HTN controlled" and have undetectable HIV viral load (at 12 months and 24 months).

SECONDARY OUTCOMES:
Lowered blood pressure | 24 months
  Proportion of HTN patients with successfully lowered BP (by at least 10 mmHg systolic and/or diastolic) compared to the time at the first HTN diagnosis
Routine Hypertension care | 12 and 24 months
  Proportion of health facilities providing hypertension care as routine practice;
Adoption of the integrated model | 12 and 24 months
  Proportion of HC IIIs and IVs adopting the integrated HIV/HTN care model;
Knowledge of HTN management and HTN complications among health workers | 12 and 24 months
  Knowledge of HTN management and complications among health workers (measured through conducting surveys among health workers working in the HIV clinics using a standardised knowledge test)
Patient satisfaction | 12 and 24 months
  Patient satisfaction outcomes in a sub-sample of facilities (survey)
Adoption of HMIS tools | 24 months
  Adoption of the integrated HIV/HTN HMIS tools particularly NCD registers and NCD patient card approved by the MoH
Service readiness for delivering hypertension care | 24 months
  Proportion of health facilities (HFs) that demonstrate service readiness for delivering adequate hypertension care for patients with and without HIV-infection
Adherence to national guidelines | 24 months
  Proportion of hypertensive patients (HIV-positive and -negative) registered at HFs that are being managed according to national guidelines.
Cost effectiveness of the integrated HIV/HTN care model | 24 months
  Incremental costs of the intervention (will be measured using micro-costing through interviews with coordinators, site visits and time-and-motion studies with clinic

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kabami, MPH, Principal Investigator — Infectious Diseases Research Collaboration, Uganda; Moses R Kamya, PhD, Principal Investigator — Infectious Diseases Research Collaboration, Uganda; Heiner Grosskurth, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: Yes
IDRC will use its proprietary Data Management system to manage and store the data throughout the life of the project. Data is transferred to the system from remote sites via an encrypted link using secure File Transfer Protocol. The system includes a data repository specific to this study which is accessible only to designated study personnel. Study staff will access the repository via a password protected website and the data will be transferred over an encrypted connection via secure Hypertext Transfer Protocol.
  After the study, clean study datasets will be made shareable in a public certified repository that supports open access. Prior to release, all datasets will be reviewed to ensure they are properly de identified. Any workflows will be exactly described and documented such that it will allow any external groups to precisely reproduce results from the raw data. IDRC will also keep the raw data on the IDRC servers for at least 5 years after the end of the study.
Time Frame: During the study and at least 5 years after the end of the study
Access Criteria: All final, clean study datasets will be made shareable in a public certified repository that supports open access.

REFERENCES:
- [Derived] Atukunda M, Kabami J, Mutungi G, Twinamatsiko B, Nangendo J, Shade SB, Charlebois E, Grosskurth H, Kamya M, Okello E. Rationale and design of leveraging the HIV platform for hypertension control in Africa: protocol of a cluster-randomised controlled trial in Uganda. BMJ Open. 2022 Dec 8;12(12):e063227. doi: 10.1136/bmjopen-2022-063227. PMID 36600388